CLINICAL TRIAL: NCT05471024
Title: Intraoral Occlusal Adjustment Time and Volume Required for Single Unit Fixed Prosthesis Fabricated With Different Virtual Articulator Mounting Methods (a Randomized Controlled Clinical Trial)
Brief Title: Occlusal Adjustment Time and Volume for Single Unit Fixed Prosthesis Fabricated With Different Virtual Mounting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aly Ayman Mohamed El-Kady, Assistant Lecturer of fixed prosthodontics, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KADY0001
Record Dates: First submitted 2022-06-28; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Dental Occlusion; Crowns
Keywords: Occlusion; Occlusal Adjustment; Virtual Articulator; Occlusal Design; Occlusal Interference
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: Triple blind (participant, investigator and outcomes assessor), randomized, clinical superiority trial with 1:1:1 allocation ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All conventional and digital mounting procedures will be performed with all trial participants and the allocation will occur as to which mounting procedure will be utilized in the designing of the crown. Sequence allocation will be performed using a random sequence generated by an impartial third party who will assign an equal number of participants to each mounting condition. This allocation will be shared with the laboratory technician but not the main investigator as he will be performing the outcomes assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digitized Mounted Articulator Scan (Active Comparator): Conventional articulator facebow mounting will be digitized using extraoral digital 3d scanner and used to position the maxillary cast on the virtual articulator.
  This positioning will be utilized during design of the occlusal surface of the restoration.
  Interventions: Procedure: Digitized Mounted Articulator Scan
- Average Positioning on Virtual Bonwill Triangle (Experimental): Virtual Bonwill triangle will be used to position the maxillary cast on the virtual articulator.
  This positioning will be utilized during design of the occlusal surface of the restoration.
  Interventions: Procedure: Average Positioning on Virtual Bonwill Triangle
- Digital Face Scan (Experimental): Digital face scan will be used to position the maxillary cast on the virtual articulator.
  This positioning will be utilized during design of the occlusal surface of the restoration.
  Interventions: Procedure: Digital Face Scan

INTERVENTIONS:
Procedure: Digitized Mounted Articulator Scan — Conventional articulator facebow mounting will be digitized using extraoral digital 3d scanner and used to position the maxillary cast on the virtual articulator. This positioning will be utilized during design of the occlusal surface of the restoration.
  Arms: Digitized Mounted Articulator Scan
Procedure: Average Positioning on Virtual Bonwill Triangle — Virtual Bonwill triangle will be used to position the maxillary cast on the virtual articulator.
  This positioning will be utilized during design of the occlusal surface of the restoration.
  Arms: Average Positioning on Virtual Bonwill Triangle
Procedure: Digital Face Scan — Digital face scan will be used to position the maxillary cast on the virtual articulator.
  This positioning will be utilized during design of the occlusal surface of the restoration.
  Arms: Digital Face Scan

SUMMARY:
Regardless of the fabrication workflow occlusal adjustments seem to be inevitable during delivery of indirect fabrication of the restoration. This has been attributed to snowballing of discrepancies due to multiple procedures for information transfer between the clinician and the laboratory. Current digital workflows minimize these discrepancies due to digital acquisition technology which eliminates drawbacks from physical materials which would alter the dimensions and morphology of the final restoration. Utilizing 3D face scanning technology is by far the least invasive and the least time consuming of available virtual facebow techniques and thus it's utilization could offer the benefit of saving time during occlusal adjustment and enhanced strength of the restoration by not subjecting it to the heat generation and subsequent crack initiation which occurs during occlusal adjustment. This study aims to compare the effect of a face scan to alignment of the maxillary cast on the volume and time of occlusal adjustment compared to conventional articulator digitization to align the maxillary cast.

DETAILED DESCRIPTION:
This study will be carried out on participants enrolled at the outpatient fixed prosthodontics clinic, Faculty of Dentistry, Cairo University.

Digital face scanning technology has made it possible to align the maxillary cast in a virtual articulator to represent a more accurate relationship to the terminal hinge axis of the patient than average positioning on a virtual Bonwill triangle. This would be reflected on the occlusal design of the restoration and subsequently on the amount of adjustment needed to the occlusal surface of the restoration during delivery. Decreasing the amount and time of occlusal adjustment would result in a decrease in chair time, increase in the longevity of the restoration and enhanced esthetics of the restoration.

Conventional alignment and mounting of casts to simulate the patients' dynamic occlusions remains the gold standard to which newer digital cast alignment and relation technology is to be compared. Thus the selection of the articulator scan as the comparator was made

Participants' Timeline

Clinical Visit 1 Preoperative records Clinical examination, Radiographic examination, Assessment of inclusion, Informed consent, Intraoral photographs, Primary impression (irreversible hydrocolloid) for diagnostic cast fabrication.

Clinical Visit 2 Facebow record, Articulator mounting, Face Scan, Foundation restoration for participant tooth built to full contour.

Clinical Visit 3 Preparation, Impression, Provisionalisation,

Allocation Impartial third party randomly allocates jaw relation methods to participants and informs laboratory technician of allocation results.

Single unit fixed prosthesis will be fabricated as per allocation results

Clinical Visit 4 Checking and verification of restoration ensuring

1. Proximal contour and contact.
2. Marginal integrity
3. Facial and lingual contours.
4. Surface finish.
5. Color and shade.

Impression prior to occlusal adjustment, Occlusal adjustment, Timing occlusal adjustment procedure, Impression after occlusal adjustment, Cementation.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 21-70 years old, be able to read and sign the informed consent document.
* Psychologically and physically able to withstand conventional dental procedures.
* Participants with molars indicated for full coverage restorations

  1. Large carious lesions
  2. Teeth restored with large restorations
  3. Endodontically treated teeth
* Accept to undergo face scanning and articulator mounting procedures
* Have no active periodontal or pulpal diseases, have teeth with clinically acceptable restorations.
* Able to attend punctually for preplanned visits and evaluation.

Exclusion Criteria:

* Participants with active resistant periodontal diseases.
* Participants with poor oral hygiene, high caries risk and uncooperative participants.
* Pregnant women.
* Participants in the growth stage with partially erupted teeth.
* Psychiatric problems or unrealistic expectations.
* Lack of opposing dentition in the area of interest.
* Restored occlusal surface opposing the planned restoration.
* The presence of a removable or fixed orthodontic appliance.
* Signs of bruxism or clenching

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-27 (Estimated)

PRIMARY OUTCOMES:
Clinical Occlusal Adjustment Time | Immediately after verification of restoration acceptability but prior to occlusal adjustment. Time will be measured until occlusal contacts of the crown have been harmonized during the delivery clinical visit.
  Time taken to harmonize occlusal contacts with participants masticatory function during delivery of the crown.Measured in minutes and seconds.

SECONDARY OUTCOMES:
Volume of Occlusal Adjustment | Before and immediately after the occlusal adjustment. Volume before occlusal adjustment - volume after occlusal adjustment of the of the crown = volume difference
  Amount of material removed from occlusal surface of restoration to harmonize occlusal contacts during delivery of the crown with participants masticatory function.

CONTACTS AND LOCATIONS:
Overall Officials: Aly AM El-Kady, MSc, Principal Investigator — Fixed Prosthodontics Department, Misr International University; Shereen A Ameen, Prof. Dr., Study Chair — Fixed Prosthodontics Department, Cairo University; Rasha NM Sami, Prof. Dr., Study Director — Fixed Prosthodontics Department, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
Only outcomes will be shared. Participants' personal information will be stored in a password protected folder.